CLINICAL TRIAL: NCT00560365
Title: A Randomised Controlled Trial to Assess the Cost-effectiveness of Intensive Versus no Scheduled Follow-up in Patients Who Have Undergone Resection for Colorectal Cancer With Curative Intent. (FACS - Follow-up After Colorectal Surgery)
Brief Title: Follow-Up Study of Patients Who Have Undergone Surgery for Stage I, Stage II, or Stage III Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000576476; USCTU-FACS; ISRCTN41458548; EU-20788
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2009-08

CONDITIONS: Colorectal Cancer
Keywords: stage I colon cancer; stage II colon cancer; stage III colon cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Magnetic Resonance Spectroscopy

INTERVENTIONS:
Other: laboratory biomarker analysis
Procedure: computed tomography
Procedure: magnetic resonance imaging
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Following patients who have undergone surgery for colorectal cancer may help doctors learn more about the disease and plan better follow-up care.

PURPOSE: This randomized clinical trial is following patients who have undergone surgery for stage I, stage II, or stage III colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the effect of augmenting symptomatic follow-up in primary care with two intensive methods of follow-up (monitoring tumor marker in primary care and intensive imaging in hospital) on survival of patients with stage I, II, or III colorectal cancer who have undergone curative resection.

Secondary

* Determine the quality of life of these patients.
* Determine the cost of National Health Service (NHS) services utilized.
* Determine the NHS cost per life-year saved.

OUTLINE: This is a multicenter study. Patients are stratified according to certainty of need for imaging follow-up, as determined by the local clinician (uncertain vs certain). Patients are randomized to 1 of 4 follow-up arms.

* Arm I (primary care follow-up): Patients undergo symptomatic follow-up (i.e., are asked to contact their physician if they have symptoms suggestive of disease recurrence). Some patients may also undergo a single CT scan 12-18 months post-randomization.
* Arm II (primary care follow-up): Patients undergo tumor marker measurements (CEA) at baseline, every 3 months for 2 years, and every 6 months for 3 years. Some patients may also undergo a single CT scan 12-18 months post-randomization.
* Arm III (intensive hospital follow-up): Patients undergo CT scan or MRI at baseline, every 6 months for 2 years, and then annually for 3 years.
* Arm IV (primary care and intensive hospital follow-up): Patients undergo primary care and intensive hospital follow-up as in arms II (without the single CT scan) and III.

All patients receive a handbook from their physician detailing possible symptoms suggestive of disease recurrence.

Quality of life is assessed at baseline and then annually for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of primary colorectal cancer

  * Stage I-III disease
* Have undergone curative resection (i.e., no residual disease [R0])

  * Microscopically clear margins
* Complete normal colonic imaging pre-operatively (or post-operatively if unable to view complete colon pre-operatively) by colonoscopy, barium enema, CT pneumocolon, or virtual colonoscopy
* Post-operative blood CEA ≤ 10 ng/mL (if the normal range is ≤ 5 ng/mL) OR < 2 times upper limit of normal (if normal range is > 5 ng/mL)

  * For patients undergoing adjuvant therapy, CEA should be measured after completion of chemotherapy
* Has completed primary curative treatment, as deemed by hospital clinician

  * Patients awaiting stoma closure allowed
* No evidence of metastatic disease on pre- or post-operative liver CT scan (or ultrasound) and chest CT scan (or chest x-ray)
* No diagnosis of familial adenomatous polyposis (FAP) or dominantly inherited colon cancer

PATIENT CHARACTERISTICS:

* No concurrent serious illness
* History of other carcinoma allowed provided primary treatment has been completed, there is no evidence of recurrent disease, and there is no follow-up that conflicts with study follow-up

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Pre-operative radiotherapy or chemoradiotherapy for rectal cancer allowed provided curative resection has been achieved
* No concurrent participation in a primary treatment clinical trial with conflicting follow-up requirements

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4760 (Estimated)
Dates: Start 2004-03; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival by intention-to-treat analysis

SECONDARY OUTCOMES:
Quality of life
Cost of National Health Service (NHS) services utilized
NHS cost per life-year saved

CONTACTS AND LOCATIONS:
Overall Officials: John N. Primrose, MD, Study Chair — University Hospital Southampton NHS Foundation Trust
Locations (31):
- United Kingdom (31):
  - Queen's Hospital, Burton-on-Trent, England
  - Cumberland Infirmary, Carlisle, England
  - Saint Richards Hospital, Chichester, England
  - Queen Alexandra Hospital, Cosham, England
  - Castle Hill Hospital, Cottingham, England
  - Mid Cheshire Hospitals Trust- Leighton Hopsital, Crewe, England
  - Mayday University Hospital, Croydon, England
  - Darent Valley Hospital, Dartford Kent, England
  - Royal Derby Hospital, Derby, England
  - Russells Hall Hospital, Dudley, England
  - Grantham and District Hospital, Grantham, Lincolnshire, England
  - Harrogate District Hospital, Harrogate, England
  - St. Mark's Hospital, Harrow, England
  - Wycombe General Hospital, High Wycombe, England
  - Hinchingbrooke Hospital, Huntingdon, England
  - West Middlesex University Hospital, Isleworth, England
  - Leeds General Infirmary, Leeds, England
  - Charing Cross Hospital, London, England
  - Mid Kent Oncology Centre at Maidstone Hospital, Maidstone, England
  - Queen's Medical Centre, Nottingham, England
  - Derriford Hospital, Plymouth, England
  - Scarborough General Hospital, Scarborough, England
  - Royal Shrewsbury Hospital, Shrewsbury, England
  - Wexham Park Hospital, Slough, Berkshire, England
  - Solihull Hospital, Solihull, England
  - Southampton General Hospital, Southampton, England
  - St. Peter's Hospital, Surrey, England
  - Royal Cornwall Hospital, Truro, Cornwall, England
  - Hillingdon Hospital, Uxbridge, England
  - Warrington Hospital NHS Trust, Warrington, England
  - Worcester Royal Hospital, Worcester, England